CLINICAL TRIAL: NCT02918773
Title: Pediatric Emergency Department Smartphone Otoscope Study (PED-Oto)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other); Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Andi L. Shane, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00090777
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Acute Otitis Media; Acute Otitis Externa
Keywords: Pediatrics; Emergency Medicine; Ear infection
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone otoscope (Experimental): Participating clinicians randomized to the smartphone otoscope study arm will use a smartphone otoscope for all otic (ear) examinations for a 6-month period.
  Interventions: Device: Smartphone otoscope
- Conventional otoscope (Active Comparator): Participating clinicians randomized to the conventional otoscope study arm will use a conventional otoscope for all otic (ear) examinations for a 6-month period.
  Interventions: Device: Conventional otoscope

INTERVENTIONS:
Device: Smartphone otoscope — A smartphone otoscope is a pocket size smartphone attachment that uses the technology and light source of a smartphone to capture reproducible images of the ear canal and tympanic membrane. The smartphone otoscope has the capability to capture still images and video, which can be referred to post-examination as well as be incorporated into an electronic medical record. Clinicians will use the smartphone otoscope for the duration of the 6-month study period.
  Other Names: CellScope-Oto
  Arms: Smartphone otoscope
Device: Conventional otoscope — A conventional otoscope has a light and lenses to provide a view of the ear canal and tympanic membrane or eardrum. Clinicians will use the conventional otoscope for the duration of the 6-month study period.
  Arms: Conventional otoscope

SUMMARY:
Acute otitis media (AOM), defined as acute inflammation in the middle ear, is a leading cause of health encounters and antimicrobial prescriptions in children worldwide. Diagnosis of AOM is often dependent on a brief view of the tympanic membrane in an uncooperative child's ear canal. As a consequence, AOM may be inappropriately diagnosed when visualization of the tympanic membrane (ear drum) is not optimal. Improved methods for visualizing the tympanic membrane including capturing still images and recording video of the ear exam would be beneficial in the diagnosis and management of otic complaints, including acute and chronic otitis media. Use of a smartphone otoscope has the potential to optimize clinician ability to manage otic complaints, visualize the tympanic membrane, and support antimicrobial stewardship. This study will be conducted as a randomized control study in two affiliated children's hospital emergency departments. Twenty volunteer clinicians will be randomly assigned to use either a smartphone otoscope or a conventional otoscope for all otic examinations for a 6-month period.

DETAILED DESCRIPTION:
A smartphone otoscope (CellScope-Oto) is a pocket size attachment that employs the technology and light source of a smartphone to capture reproducible images of the ear canal and tympanic membrane. Previous studies with this device demonstrated that images taken with both the smartphone otoscope and a camera-fitted conventional analogue otoscope were equivalent with respect to image quality and that the smartphone otoscope was acceptable as an educational and diagnostic tool to health professional students. A pilot study with a similar design to this study conducted in two offices of an ambulatory pediatric clinic demonstrated a trend toward decreased antimicrobial prescription filling among families whose children were examined with the smartphone otoscope compared to those who were examined with a conventional otoscope. To further assess this trend, this study proposes an evaluation of the impact of device use on antimicrobial prescribing for children with an otic complaint in a pediatric emergency department (PED) setting. This study will enroll 20 clinicians for the 6-month study period; 10 who will be randomly assigned to use a smartphone otoscope for the 6-month study period and 10 who will be assigned to use a conventional otoscope for all otoscopic exams. Data will be abstracted via retrospective review of the electronic medical record of encounters in with an otoscopic exam was performed as part of the diagnostic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a pediatric emergency care clinicians providing care at an emergency department a participating children's hospital
* Willing to agree to random assignment to either a smartphone otoscope device or a conventional otoscope device for the 6-month study period
* Willing to log patient encounters that included the an otoscopic examination for non-traumatic indication for each shift
* Willing to document and report episodes of care in which the assigned otoscopic device could not be used on a study-eligible otoscopic examination
* Willing to complete an end of study assessment, if assigned to use the smartphone otoscope

Exclusion Criteria:

* Declines to give informed consent to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Shane, MD, MPH, MSc, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta at Hughes Spalding, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-two volunteer clinicians were randomly assigned to use either a smartphone otoscope device or a conventional otoscope for a six-month period from October 15, 2016 to April 15, 2017. This study was conducted at two children's hospital emergency departments in Atlanta, Georgia.
Pre-assignment Details: Study clinicians logged 1,502 encounters where otoscopes were used; 112 (7%) of encounters were excluded due to incomplete data or not meeting study inclusion criteria, for a total of 1390 encounters evaluated.
Units Other Than Participants: Emergency department encounters
Groups:
- Conventional Otoscope Encounters: Emergency department encounters by participating clinicians randomized to the conventional otoscope study arm. Clinicians randomized to this group used a conventional otoscope for a 6-month period for all otic (ear) examinations for any non-traumatic complaints with the potential for otic involvement including fever, ear pain, congestion, or runny nose.
- Smartphone Otoscope Encounters: Emergency department encounters by participating clinicians randomized to the smartphone otoscope study arm. Clinicians randomized to this group used a smartphone otoscope for a 6-month period for all otic (ear) examinations for any non-traumatic complaints with the potential for otic involvement including fever, ear pain, congestion, or runny nose.
Period: Overall Study
Arm/Group | Conventional Otoscope Encounters | Smartphone Otoscope Encounters
Started | 11; 776 Emergency department encounters | 11; 614 Emergency department encounters
Completed | 11; 776 Emergency department encounters | 11; 614 Emergency department encounters
Not Completed | 0; 0 Emergency department encounters | 0; 0 Emergency department encounters

BASELINE CHARACTERISTICS:
Population: The attributes of the children seen in the pediatric emergency department who were examined by clinicians participating in the study are presented in the baseline analysis. Only minimal information was collected from the medical records regarding the baseline characteristics of these children..
Units Other Than Participants: ED encounters
Groups:
- Conventional Otoscope Encounters: Emergency department (ED) encounters by participating clinicians randomized to the conventional otoscope study arm. Clinicians randomized to this group used a conventional otoscope for a 6-month period for all otic (ear) examinations for any non-traumatic complaints with the potential for otic involvement including fever, ear pain, congestion, or runny nose.
- Smartphone Otoscope Encounters: Emergency department (ED) encounters by participating clinicians randomized to the smartphone otoscope study arm. Clinicians randomized to this group used a smartphone otoscope for a 6-month period for all otic (ear) examinations for any non-traumatic complaints with the potential for otic involvement including fever, ear pain, congestion, or runny nose.
- Total: Total of all reporting groups
Arm/Group | Conventional Otoscope Encounters | Smartphone Otoscope Encounters | Total
Number analyzed (Participants) | 11 | 11 | 22
Number analyzed (ED encounters) | 776 | 614 | 1390
Age, Continuous [Mean (Standard Deviation); unit: age in months of encounter subjects] — Population: The age of one child in the smartphone otoscope group is unknown.
  age in months of encounter subjects
    number analyzed (ED encounters) | 776 | 613 | 1389
    (all) | 43.5 (38.8) | 49.0 (42.0) | 45.90 (40.34)
Sex/Gender, Customized [Number; unit: Emergency department encounters]
  Not collected | 776 | 614 | 1390
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: Emergency department encounters]
  United States | 776 | 614 | 1390
Reason for clinic visit [Number; unit: Emergency department encounters] — A child could have multiple symptoms documented as the reason for the emergency department visit.
  Emergency department encounters
    Fever | 522 | 424 | 946
    Ear pain | 106 | 96 | 202
    Congestion/runny nose | 270 | 182 | 452
    Cough | 365 | 274 | 639
    Other | 338 | 317 | 655

OUTCOME MEASURES:

1. Primary Outcome: Number of Antibiotic Prescriptions
Description: The number of emergency department encounters where antibiotics were prescribed to treat acute otitis media (AOM) are presented here. Information about antimicrobial prescriptions were found in the medical records of children receiving an otoscopic exam by a participating clinician.
Time Frame: Month 6
Population: This analysis includes emergency department encounters with children by a participating clinician where AOM was diagnosed.
Measure: Number; unit: Emergency department encounters
Units Other Than Participants: Number of encounters
Arm/Group | Conventional Otoscope Encounters | Smartphone Otoscope Encounters
Number analyzed (Participants) | 11 | 11
Number analyzed (Number of encounters) | 146 | 123
Emergency department encounters
  Antibiotic prescribed | 140 | 115
  Antibiotic not prescribed | 6 | 7
  Unknown | 0 | 1

2. Secondary Outcome: Number of Diagnoses of Acute Otitis Media (AOM)
Description: The number of emergency department encounters where a diagnosis of acute otitis media (AOM) was made is presented here. Information about the diagnosis of AOM was found in the medical records of children receiving an otoscopic exam by a participating clinician.
Time Frame: Month 6
Measure: Number; unit: Emergency department encounters
Units Other Than Participants: Clinic encounters
Arm/Group | Conventional Otoscope Encounters | Smartphone Otoscope Encounters
Number analyzed (Participants) | 11 | 11
Number analyzed (Clinic encounters) | 776 | 614
Emergency department encounters
  AOM Diagnosed | 146 | 123
  AOM Not Diagnosed | 630 | 491

3. Secondary Outcome: Number of Diagnoses of Otitis Externa
Description: The number of emergency department encounters where a diagnosis of otitis externa was made is presented here. Information about the diagnosis of otitis externa was found in the medical records of children receiving an otoscopic exam by a participating clinician.
Time Frame: Month 6
Measure: Number; unit: Emergency department encounters
Units Other Than Participants: Clinic encounters
Arm/Group | Conventional Otoscope Encounters | Smartphone Otoscope Encounters
Number analyzed (Participants) | 11 | 11
Number analyzed (Clinic encounters) | 776 | 614
Emergency department encounters
  Otitis Externa Diagnosed | 0 | 0
  Otitis Externa Not Diagnosed | 776 | 614

4. Secondary Outcome: Clinician Acceptability of the Smartphone Otoscopic Device
Description: Clinicians randomized to use the smartphone otoscopic device completed a survey to assess the acceptability of this device compared to the historical use of a conventional otoscope. The survey, developed specifically for this study, asked clinicians to report on their preference for using the smartphone otoscope over the conventional otoscope, whether the device increased their ability to diagnose AOM, and the perceived impact on antibiotic prescribing.
Time Frame: Month 6
Population: Only participating clinicians who were randomized to use the smartphone otoscope were administered a survey at the end of the 6-month intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Clinicians Assigned to the Smartphone Otoscope Group: Clinicians assigned to this study arm used a smartphone otoscope rather than a conventional otoscope for all otic examinations during the six month intervention period.
Arm/Group | Clinicians Assigned to the Smartphone Otoscope Group
Number analyzed (Participants) | 11
Participants
  Preferred smartphone over conventional otoscope | 8
  Smartphone increased ability to diagnose AOM | 3
  Smartphone did not impact antibiotic prescribing | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 6-month intervention period of October 15, 2016 to April 15, 2017.
Description: This study collected any adverse events related to otoscope use, however, adverse events were not expected as the intervention does not pose more than minimal risk to patients being examined. Adverse events are reported on the emergency department encounter level rather than the clinician participant level.
Arm/Group | Conventional Otoscope Encounters | Smartphone Otoscope Encounters
All-Cause Mortality (participants affected / at risk) | 0/776 | 0/614
Serious Adverse Events (participants affected / at risk) | 0/776 | 0/614
Other Adverse Events (participants affected / at risk) | 0/776 | 0/614

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02918773/Prot_SAP_000.pdf